CLINICAL TRIAL: NCT03616002
Title: Effects of Hookah Smoking on Vascular Regulation: Novel Insight Into Endothelial Function
Brief Title: Effects of Hookah (Waterpipe) Smoking on Blood Vessel Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due tot he Pandemic we decided to terminate this project.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Los Angeles (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Florian Rader, M.D, M.Sc., Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00036547
Record Dates: First submitted 2015-01-13; First posted 2018-08-06 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hookah Smoking
MeSH Terms: conditions — Water Pipe Smoking | interventions — Smoking Water Pipes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hookah smoking (Experimental): Healthy habitual Hookah smokers will undergo brachial artery flow mediated dilation, reactive hyperemia peripheral arterial tonometry or pulse tonometry before and after Hookah smoking.
  Interventions: Other: Hookah smoking

INTERVENTIONS:
Other: Hookah smoking — ad lib hookah smoking for 30 minutes in a controlled laboratory environment.

SUMMARY:
The purpose of this study is to assess the acute effects of Hookah (waterpipe) smoking on blood vessel function. Hookah smoking has been shown to immediately increase blood pressure and heart rate which could result in damage in the inner lining of the body's blood vessels.

DETAILED DESCRIPTION:
The investigators will measure acute endothelial and vascular changes before and after a 30-minute Hookah smoking session in a controlled laboratory environment to: (1) Determine the acute effects of Hookah smoking on large-vessel endothelial vasodilator function measured by brachial artery flow mediated dilation; (2) Determine the acute effects of Hookah smoking on micro-vessel endothelial function as measured by reactive hyperemia peripheral arterial tonometry; (3) Determine the acute effects of Hookah smoking on pulse wave velocity and aortic pressure waveform measured by pulse tonometry.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 29 years of age
* Habitual Hookah smoker defined as having smoked Hookah >=12 times in the past 12 months
* Have not smoked cigarettes within the past 12 months

Exclusion Criteria:

* History of cardiopulmonary, diabetes, dyslipidemia or psychiatric disease
* Exhaled carbon monoxide level >10 ppm
* BP < 140/90 mmHg
* BMI <18.5 or > 30 kg•m2
* Resting heart rate > 100 beats/min
* Taking prescription medication
* History of illicit drug use
* Pregnant

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | change from baseline to immediately after smoking

SECONDARY OUTCOMES:
Reactive hyperemia peripheral arterial tonometry | change from baseline to immediately after smoking

OTHER OUTCOMES:
Pulse wave velocity | change from baseline to immediately after smoking
aortic pressure waveform | change from baseline to immediately after smoking

CONTACTS AND LOCATIONS:
Overall Officials: Florian Rader, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezk-Hanna M, Mosenifar Z, Benowitz NL, Rader F, Rashid M, Davoren K, Moy NB, Doering L, Robbins W, Sarna L, Li N, Chang LC, Elashoff RM, Victor RG. High Carbon Monoxide Levels from Charcoal Combustion Mask Acute Endothelial Dysfunction Induced by Hookah (Waterpipe) Smoking in Young Adults. Circulation. 2019 May 7;139(19):2215-2224. doi: 10.1161/CIRCULATIONAHA.118.037375. PMID 30764644